CLINICAL TRIAL: NCT06278090
Title: Impact of Ursodeoxycholic Acid Treatment on the Gallbladder Polyp Evolution. Prospective Cohort Study
Brief Title: Impact of Ursodeoxycholic Acid Treatment on the Gallbladder Polyp Evolution
Acronym: GALPOL
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Tihomir Georgiev Hristov, Principal Investigator, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Other Study IDs: AUDC
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Gallbladder Polyp
Keywords: Gallbladder polyp; Ursodeoxycholic acid
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with Ursodeoxycholic acid: Patients that recieved prescription for Ursodeoxycholic acid, 10-15 mg/kg for at least 6 months.
  Interventions: Drug: Ursodeoxycholic Acid Only Product
- Patients not treated with Ursodeoxycholic acid: Patients without prescription of Ursodeoxycholic acid

INTERVENTIONS:
Drug: Ursodeoxycholic Acid Only Product — Ursodeoxycholic acid treatment, 10-15mg/kg/day for at least 6 months
  Other Names: Ursobilane, Ursochol
  Groups: Patients treated with Ursodeoxycholic acid

SUMMARY:
The goal of this observational study is to learn about the impact of ursodeoxycholic acid treatment on the gallbladder polyp evolution in patients with gallbladder polyps that undergo follow up. The main question it aims to answer is:

• Whether ursodeoxycholic acid could decrease the gallbladder polyp size and therefore spare unnecessary follow up or surgical interventions

Participants will be managed according to the standard practice of the department they are attended:

* According to the established practice in the Department of Surgery, patients that either do not have an indication for cholecystectomy or decline the offered intervention, and are subjects for a follow up, are usually prescribed Ursodeoxycholic Acid, at 10-15 mg/kg/day for at least 6 months.
* According to the standard practice of Gastroenterology Department, patients are followed up according to the published guidelines.

Researchers will compare the groups that receive or not ursodeoxycolic acid treatment to see if the polyp size evolution differs significantly.

DETAILED DESCRIPTION:
Gallbladder polyps are common findings on abdominal ultrasound studies. Most of them are cholesterol polyps. However, often they require a prolonged follow up due to impossibility to efficiently rule out the presence of a real adenomatous polyps with potential of malignization.

Ursodeoxycholic Acid is a well-studied and long known drug that has been used for conservative treatment of bile stones with high cholesterol concentration (most of them), but also for bile sludge and gallbladder polyps, that are considered precursors of the gallbladder stones. It has been found in several studies that prevent from recurrent idiopathic acute pancreatitis and from gallbladder stone formation after gastric (including bariatric) surgery.

Participants will be managed according to the standard practice of the department they are attended:

* According to the established practice in the Department of Surgery, patients that either do not have an indication for cholecystectomy or decline the offered intervention, and are subjects for a follow up, are usually prescribed ursodeoxycholic acid, at 10-15 mg/kg/day for at least 6 months.
* According to the standard practice of Gastroenterology Department, patients are followed up according to the published guidelines.

Researchers will compare the groups that receive or not ursodeoxycolic acid treatment to see if the polyp size evolution differ significantly during the studied period of 1 year. The small size changes could have a great impact on the management of the gallbladder polyps as for a 2mm increase could be a reason to indicate a surgical intervention and a 2mm decrease could cause the discontinuation of the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gallbladder polyps eligible for standard follow up (without indication for cholecystectomy or patient decline surgery or polyps < 5mm without risk factors such as age>60 years, primary sclerosing cholangitis, asian ethnicity, sessile polypoid lesion)

Exclusion Criteria:

* Patients with gallbladder polyps that received ursodeoxycolic acid doses lower than 10mg/kg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred for an outpatient consultation to the Departments of Surgery and Gastroenterology due to gallbladder polyps.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Reducing gallbladder polyp size by 2mm or more | 6 and 12 months
  Reducing the polyp size by 2mm or more, at the usual ultrasonographic controls at 6 and 12 months.

SECONDARY OUTCOMES:
Modification of the expected follow up | 12 months
  Depending on the polyp size, physicians could either discontinue the follow up (decreasing to <5mm or disappearing) or indicate surgery (according to the current guidelines). Deviation from the usual evolution of the polyp size, comparing both groups, that leads to alteration of the possible follow up (termination of the follow up when polyp size reduces to <5mm or indication of surgery when polyp size increases by 2mm or reaches 10mm) will be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Tihomir Georgiev, MD, PhD, Principal Investigator — Hospital Universitario General de Villalba, Madrid, Spain
Locations (1):
- Hospital Universitario General de Villalba, Collado Villalba, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No